CLINICAL TRIAL: NCT00782717
Title: A Clinical Safety and Efficacy Comparison of NEVANAC 0.1% to Vehicle Following Cataract Surgery in Diabetic Retinopathy Patients
Brief Title: A Clinical Safety and Efficacy Comparison of NEVANAC 0.1% to Vehicle After Cataract Surgery in Diabetic Retinopathy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C-07-43
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2011-09-21 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Macular Edema
Keywords: diabetic retinopathy; cystoid macular edema;
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy | interventions — nepafenac; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEVANAC (Experimental): One drop three times a day starting on the day prior to cataract surgery (Day -1) and continuing on the day of surgery (Day 0) and for 90 days thereafter.
  Interventions: Drug: Nepafenac ophthalmic suspension, 0.1% (NEVANAC); Drug: Prednisolone acetate ophthalmic suspension (OMNIPRED)
- Nepafenac Vehicle (Placebo Comparator): One drop three times a day starting on the day prior to cataract surgery (Day -1) and continuing on the day of surgery (Day 0) and for 90 days thereafter.
  Interventions: Other: Nepafenac ophthalmic suspension vehicle; Drug: Prednisolone acetate ophthalmic suspension (OMNIPRED)

INTERVENTIONS:
Drug: Nepafenac ophthalmic suspension, 0.1% (NEVANAC) — 1 drop TID beginning the day before surgery, continuing on the day of surgery and through the first 90 days following surgery.
  Other Names: NEVANAC
  Arms: NEVANAC
Other: Nepafenac ophthalmic suspension vehicle — 1 drop TID beginning the day before surgery, continuing on the day of surgery and through the first 90 days following surgery
  Arms: Nepafenac Vehicle
Drug: Prednisolone acetate ophthalmic suspension (OMNIPRED) — One drop in the study eye 4 times daily (morning, late morning, late afternoon, and bedtime)for two weeks postsurgery.
  Other Names: OMNIPRED

SUMMARY:
The purpose of this study is to determine whether nepafenac is safe and effective for reducing the incidence of macular edema following cataract surgery in diabetic retinopathy patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-proliferative diabetic retinopathy (mild, moderate or severe) and planned cataract extraction by phacoemulsification.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Central subfiled macular thickness greater than or equal to 250 microns
* CME in either eye.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

REFERENCES:
- [Result] Singh R, Alpern L, Jaffe GJ, Lehmann RP, Lim J, Reiser HJ, Sall K, Walters T, Sager D. Evaluation of nepafenac in prevention of macular edema following cataract surgery in patients with diabetic retinopathy. Clin Ophthalmol. 2012;6:1259-69. doi: 10.2147/OPTH.S31902. Epub 2012 Aug 3. PMID 22927737
- [Derived] Pollack A, Staurenghi G, Sager D, Mukesh B, Reiser H, Singh RP. Prospective randomised clinical trial to evaluate the safety and efficacy of nepafenac 0.1% treatment for the prevention of macular oedema associated with cataract surgery in patients with diabetic retinopathy. Br J Ophthalmol. 2017 Apr;101(4):423-427. doi: 10.1136/bjophthalmol-2016-308617. Epub 2016 Jul 7. PMID 27388251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 41 investigative centers from November 2008 to July 2010. 263 patients diagnosed with diabetic retinopathy and requiring cataract extraction with intraocular lens implantation were randomized.
Pre-assignment Details: Of the 263 patients enrolled, 12 exited prior to surgery. Baseline characteristics are presented for the ITT population, i.e., patients who were exposed to the study drug, completed the implant surgery, and had at least one on-therapy post-surgical visit.
Period: Overall Study
Arm/Group | NEVANAC | Nepafenac Vehicle
Started | 133 | 130
Completed | 118 | 102
Not Completed | 15 | 28
Not completed — Adverse Event | 2 | 5
Not completed — Patient decision unrelated to AE | 6 | 3
Not completed — Noncompliance | 2 | 1
Not completed — Treatment failure | 3 | 14
Not completed — Enrollment close prior to surgery | 1 | 0
Not completed — Did not meet entrance criteria | 1 | 3
Not completed — Exited in error | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NEVANAC | Nepafenac Vehicle | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 54 | 100
  >=65 years | 79 | 72 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 75 | 158
  Male | 42 | 51 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Developed Macular Edema (ME) Within 90 Days Following Cataract Surgery
Description: Macular edema (thickening of the center of the back of the eye) was defined as 30% or greater increase from pre-operative baseline measurement in central subfield macular thickness as measured using Optical Coherence Tomography(OCT).
Time Frame: 3 Months
Population: All patients who were exposed to the study drug, completed the implant surgery, and had at least one on-therapy post-surgical visit at which optical coherence tomography (OCT) was performed (ITT).
Measure: Number; unit: Percentage of patients
Arm/Group | NEVANAC | Nepafenac Vehicle
Number analyzed (Participants) | 125 | 126
Percentage of patients | 3 | 17

2. Secondary Outcome: Percent of Patients With a Decrease of More Than 5 Letters in Best-corrected Visual Acuity (BCVA).
Description: BCVA was measured using the procedure developed for the Early Treatment Diabetic Retinopathy Study.
Time Frame: From Day 7 to Day 90 (or Early Exit)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | NEVANAC | Nepafenac Vehicle
Number analyzed (Participants) | 124 | 122
Percentage of patients | 6 | 12

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 04 NOV 2008 to 15 JUL 2010.
Description: The safety population included all patients who received exposure or potential exposure to the study drug.
Arm/Group | NEVANAC | Nepafenac Vehicle
Serious Adverse Events (participants affected / at risk) | 4/126 | 9/127
Other Adverse Events (participants affected / at risk) | 9/126 | 19/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NEVANAC (N=126) | Nepafenac Vehicle (N=127)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Device failure (General disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Labyrnthitis (Infections and infestations) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NEVANAC (N=126) | Nepafenac Vehicle (N=127)
Eye Pain (Eye disorders) | 1 (1) | 3 (3)
Eye inflammation (Eye disorders) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review study related information prior to presentation or publication